CLINICAL TRIAL: NCT05697913
Title: Efficacy of Response-adapted Treatment Guided by Negative Minimal Residual Disease and Negative Imaging (MRDI) in Fit Patients Diagnosed With Multiple Myeloma Who Are Candidates for Bone Marrow Transplantation
Brief Title: Efficacy of Response-adapted Treatment in Patients With Multiple Myeloma Candidates for Bone Marrow Transplantation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Responsible Party: Principal Investigator, Jose Enrique de la Puerta, MD, Principal Investigator, Hospital Galdakao-Usansolo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRD-Image neg 01
Record Dates: First submitted 2022-12-25; First posted 2023-01-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma
Keywords: Minimal Residual Disease; Therapeutics; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual

STUDY DESIGN:
Intervention Model Description: Prospective, no randomized. It is a cohort study to compare MRDI(-) driven treatment adapted to the response versus fixed-duration therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRDI-driven treatment (Experimental): Patients continue treatment until complete remission with negative MRD and Image is achieved, changing the therapeutic line if this is not achieved with the prescribed treatment. In this group of patients, treatment is suspended only when this degree of profound response is reached, in any phase of treatment.
  Interventions: Other: Continued treatment adapted to the response
- Conventional treatment (No Intervention): The patients of the conventional treatment group (control group) received six cycles of the induction traetment, bone marrow auto-transplantation, and consolidation treatment after transplantation if complete remission had not been achieved.

INTERVENTIONS:
Other: Continued treatment adapted to the response — Instead of receiving a pre-specified number of treatment cycles, regardless of the result obtained, in the MRDI-driven treatment group patients continue receiving treatment until reaching a complete remission with negative MRD and Image, changing the therapeutic line if it is not obtained with the line current therapy. In this group of the patients the treatment was stopped only when this degree of deep response was achieved.
  Arms: MRDI-driven treatment

SUMMARY:
To assess whether continued treatment to achieve negative Minimal Residual Disease and Imaging (MRDI(-)) improves therapeutic outcomes in patients with newly diagnosed Multiple Myeloma. The primary endpoints are progression-free survival (PFS) and overall survival (OS). The safety evaluation includes the evaluation of adverse events, which are classified according to the Common Criteria for Terminology for Adverse Events of the National Cancer Institute, version 5.0.

DETAILED DESCRIPTION:
Material and methods - Criteria for Enrollment Patients younger than 76 years, diagnosed with myeloma since July 1, 2014 until May 31, 2019, without a contraindication for bone marrow auto-transplantation are included in the study. Fragile patients with severe senile dementia, with another non-treatable neoplasm, or with significant comorbidity in whom the therapeutic objective was only palliative are not included in the study. The allocation to each treatment group was carried out according to the patient's preferences and his/her responsible physician, giving the patient his/her consent for treatment in all cases. In addition to other information, before patients gave their consent, patients included in the continued treatment group were clarified that it was a non-standard treatment, giving them the choice between the most common option of fixed treatment or continuous treatment up to Minimal Residual Disease and Image negative (MRDI(-)).

Material and methods - Study Design and Treatment This is a study of the patients treated in real life hematology. It is a cohort study to compare continuous treatment versus fixed-duration therapy. The study is conducted in a single hospital, including patients diagnosed from July 1, 2014 to May 31, 2019. The autotransplant is considered as a therapeutic line more, and all patients who did not receive the transplant were analyzed as if they had received it. The patients always receive some of the authorized treatments for their therapeutic line, according to the preferences of the responsible hematologist and the patient. After the induction phase, all the patients undergo stem-cell mobilization with granulocyte colony-stimulating factor.

The patients of the fixed treatment group (control group) receive up to six cycles of the consolidation treatment after transplantation if complete remission has not been achieved.

In the patients of the MRDI-driven group, patients continue treatment after transplantation to achieve complete remission with negative MRD and negative image, changing therapeutic line if not achieved with the prescribed treatment. In this group of the patients the treatment is stopped only when this degree of deep response is achieved, in whatever the treatment phase was.

Assessments The treatment response and disease progression are assessed according to the International Uniform Response Criteria for Multiple Myeloma, except that to consider the negative Minimal Residual Disease, a sensitivity level of 10-6 is required. In addition, it is considered negative image only if a Positron Emission Tomography/Computed Tomography (PET/CT) body and spinal and pelvic Nuclear Magnetic Resonance (NMR), are both negative.

The work team defined an additional category of relapse: "relapse from MRDI(-)", which includes any of the relapse criteria of negative Minimal Residual Disease, and/or positive image. To evaluate the Positron Emission Tomography/Computed Tomography (PET/CT) the criteria of Elena Zamagni are used. In Nuclear Magnetic Resonance studies, all lesions with a size equal to or greater than 5 mm are considered positive if they are hypointense signal in T1, hyperintense in Fat Suppression (FS) T2 signal, and in the studies of diffusion hyperintense signal in b1000 with apparent diffusion coefficient (ADC) between 0.4 and 1. In perfusion studies, type 4-curve lesions are considered positive. The adverse events are assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 of the National Cancer Institute. It is considered as an Adverse Event (AE) any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure.

Among all the patients, bone marrow samples are obtained at diagnostic for cytogenetic evaluation.

Among the patients of the MRDI-driven group who are a complete response, bone marrow samples are obtained for minimal residual disease evaluation by means of seven-color flow cytometry (which has a sensitivity level of 10-6, indicating that it can detect 1 malignant plasma cell within 1,000,000 bone marrow cells). If the patient achieve a Complete Remission (CR) according to the International Uniform Response Criteria for Multiple Myeloma, Minimal Residual Disease (MRD) and imaging studies are performed before transplantation, after transplantation, and after every six cycles of treatment in cases with CR where previous MRD or imaging studies are positive.

In the control group, the MRD and imaging only occasionally is it evaluated. In all patients who achieve a negative MRD and negative image, MRD and imaging tests are performed at 6 months and annually.

The response obtained, progression-free survival, overall survival, and the incidence of adverse effects are valued.

Statistical Analysis Progression-free survival is defined as the time from start of treatment until either the first documentation of disease progression or death owing to myeloma or not. Overall survival is defined as the time from start of treatment until death from any cause.

Duration of PFS and OS is estimated by means of the test of the long rank Kaplan-Meier method with Cox analysis. Analyses are performed with the use of IBM SPSS Statistics software, version 23.0; the data cutoff date is June 30, 2024.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 76 years
* Diagnosed with Multiple Myeloma from July 1, 2014 to May 31, 2019
* Received some of the standard authorized treatments for their therapeutic line. Patients treated in clinical trials with treatments not yet authorized, for fifth or successive therapeutic lines are admitted.
* Give informed consent
* Fit patient

Exclusion Criteria:

* Under 18 years old
* Contraindication for bone marrow auto-transplantation
* Therapeutic objective only palliative:

  * Another non-treatable neoplasm
  * Severe senile dementia
  * Significant comorbidity limiting life expectancy to less than 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Time elapsed from start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months.
  Time elapsed from start of treatment until first documentation of disease progression or date of death from any cause, whichever came first.
Overall Survival | Time elapsed from start of treatment to end of follow-up or patient death, whichever came first, assessed up to 120 months.
  Time from start of treatment to death from any cause
Proportion of patients with serious adverse effects | Time elapsed from start of treatment to end of follow-up or patient death, whichever came first, assessed up to 102 months.
  Number of patients with any adverse event grade 3 or higher, divided by the total number of patients in the corresponding group
Average grade 3 or higher adverse events per patient | Time elapsed from start of treatment to end of follow-up or patient death, whichever came first, assessed up to 120 months.
  Number of grade 3 or higher adverse events in the group divided by the number of patients in the group
Annual incidence of grade 3 or higher adverse effects | Time elapsed from start of treatment to end of follow-up or patient death, whichever came first, assessed up to 102 months.
  Number of grade 3 or higher adverse events in the group divided by the sum of the years of observation of the group members

CONTACTS AND LOCATIONS:
Overall Officials: Jose Enrique de la Puerta Rueda, MD, Principal Investigator — Hospital Cruz Roja de Bilbao

IPD SHARING:
Plan to Share IPD: No
At this time, no plan has been developed to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Ludwig H, Zojer N. Fixed duration vs continuous therapy in multiple myeloma. Hematology Am Soc Hematol Educ Program. 2017 Dec 8;2017(1):212-222. doi: 10.1182/asheducation-2017.1.212. PMID 29222258
- [Background] Jackson GH, Davies FE, Pawlyn C, Cairns DA, Striha A, Collett C, Waterhouse A, Jones JR, Kishore B, Garg M, Williams CD, Karunanithi K, Lindsay J, Wilson JN, Jenner MW, Cook G, Kaiser MF, Drayson MT, Owen RG, Russell NH, Gregory WM, Morgan GJ; UK NCRI Haematological Oncology Clinical Studies Group. Response-adapted intensification with cyclophosphamide, bortezomib, and dexamethasone versus no intensification in patients with newly diagnosed multiple myeloma (Myeloma XI): a multicentre, open-label, randomised, phase 3 trial. Lancet Haematol. 2019 Dec;6(12):e616-e629. doi: 10.1016/S2352-3026(19)30167-X. Epub 2019 Oct 14. PMID 31624047
- [Background] Paiva B, Puig N, Cedena MT, Rosinol L, Cordon L, Vidriales MB, Burgos L, Flores-Montero J, Sanoja-Flores L, Lopez-Anglada L, Maldonado R, de la Cruz J, Gutierrez NC, Calasanz MJ, Martin-Ramos ML, Garcia-Sanz R, Martinez-Lopez J, Oriol A, Blanchard MJ, Rios R, Martin J, Martinez-Martinez R, Sureda A, Hernandez MT, de la Rubia J, Krsnik I, Moraleda JM, Palomera L, Bargay J, Van Dongen JJM, Orfao A, Mateos MV, Blade J, San-Miguel JF, Lahuerta JJ; GEM (Grupo Espanol de Mieloma)/PETHEMA (Programa Para el Estudio de la Terapeutica en Hemopatias Malignas) Cooperative Study Group. Measurable Residual Disease by Next-Generation Flow Cytometry in Multiple Myeloma. J Clin Oncol. 2020 Mar 10;38(8):784-792. doi: 10.1200/JCO.19.01231. Epub 2019 Nov 26. PMID 31770060
- [Background] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158
- [Background] Zamagni E, Nanni C, Mancuso K, Tacchetti P, Pezzi A, Pantani L, Zannetti B, Rambaldi I, Brioli A, Rocchi S, Terragna C, Martello M, Marzocchi G, Borsi E, Rizzello I, Fanti S, Cavo M. PET/CT Improves the Definition of Complete Response and Allows to Detect Otherwise Unidentifiable Skeletal Progression in Multiple Myeloma. Clin Cancer Res. 2015 Oct 1;21(19):4384-90. doi: 10.1158/1078-0432.CCR-15-0396. Epub 2015 Jun 15. PMID 26078390